CLINICAL TRIAL: NCT05292573
Title: MicroRNAs as Biomarkers of Predicting Future Endometrial Malignancy and Longitudinal Follow-up With Randomized Intervention in Women With Endometrial Hyperplasia Without Atypia
Brief Title: Longitudinal Follow-up in Women With Endometrial Hyperplasia Without Atypia
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 107-2314-B-182A-166-MY3
Record Dates: First submitted 2021-08-04; First posted 2022-03-23 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2021-07

CONDITIONS: Female
Keywords: simple hyperplasia; Metformain
MeSH Terms: interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- metformin group (Experimental): 1. During the intervention period, metformin is given 500 mg tablet b.i.d.
  2. We will deliver education for exercise and weight control to all eligible participants
  Interventions: Drug: Metformin
- Observation group (No Intervention): only exercise and weight control to all eligible participants

INTERVENTIONS:
Drug: Metformin — During the intervention period, metformin is given 500 mg tablet b.i.d. Those who stopped taking metformin will remain in the study not counting as protocol violation.
  Other Names: Uformin Tablet 500mg
  Arms: metformin group

SUMMARY:
This study will prospectively enroll a total of 1000 patients (200 per year) simple hyperplasia/complex hyperplasia (SH/CH) without atypia. All subjects will receive education for exercise and weight control and be randomized 1:1 to with or without metformin intervention. At the end of this 3-year project, an interim analysis will be performed. Since long-term follow-up is intended, therefore for the 4th to 6th year a new grant support will be looked for. The long-term occurrence of endometrial cancer (up to15 years) data will be acquired from national cancer registry, which permission is addressed in the informed sent.

DETAILED DESCRIPTION:
The first year: (1) the cumulative progression rate of SH/CH without atypia to endometrial cancer (EC) of the 1989-2011 cohort will be investigated by linking with national health databases from Health and Welfare Data Science Center (HWDC); (2) Prospectively enroll 200 patients with SH/CH without atypia and deliver education for exercise and weight control and collect the related biospecimens and data; (3) 1:1 randomized to with or without metformin intervention.

The 2nd year: (1) analyze the whole genome sequencing (WGS) data of those progressed and non-progressed ; (2) analyze the metabolomic data in relation to exercise and weight control data.

The 3rd year: (1) validate microRNA (miR) panel in tissues and sera selected by CMRPG3G1511-3; (2) analyze data of MiR panel, degree of exercise/weight control, clinical lab data, and demographic data on EC progression rate; (3) Incremental predicting proficiency of the model including metabolomics data and WGS.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged ≧ 20 years
2. Histological diagnosis of SH/CH without atypia
3. Not taking Metformin for diabetes mellitus currently
4. Adequate kidney function
5. Provided informed consent within 3 months of diagnosis
6. No previous history of breast cancer with tamoxifen use
7. Willing to be followed for 5 years

Exclusion Criteria:

1. Atypical hyperplasia or EC found within 3 months after enrollment
2. History or concurrent gynecologic cancers or cervical intraepithelial neoplasia
3. Pregnancy test positive
4. History of intolerance to Metformin
5. Family history of HNPCC

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2022-10-01 (Estimated); Study Completion 2026-01-29 (Estimated)

PRIMARY OUTCOMES:
The area under the receiver operating characteristic curve (ROC curve) (AUC) of the prediction miR panel of the 3 miRs. | 5 years
  The primary endpoint of the randomized prospective study is to evaluate the ROC of the prediction miR panel of the 3 miRs.

SECONDARY OUTCOMES:
Time to progression among groups | 3 years
  Incidence of progression to endometrial cancer among groups, Proportion of participants with treatment-related adverse events as assessed by CTCAE v4.0
Subgroup analysis in body-weight control | 3 years
  Follow up the body-weight control

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital, Linkou Branch, Taoyuan District, Taiwan